CLINICAL TRIAL: NCT06457607
Title: Prospective, Single Center, Single Arm, Open Label Study to Evaluate the Efficacy and Safety of Treatment With LinearFirm(ULTRAcel Q+) in Temporary Eyebrow Lifting
Brief Title: Evaluating the Efficacy and Safety of Treatment With LinearFirm(ULTRAcel Q+) in Temporary Eyebrow Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeisys Medical Inc (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JE_ULTRA_P01
Record Dates: First submitted 2024-06-02; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: High Intensity Focused Ultrasound
Keywords: High Intensity Focused Ultrasound; Lifting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm is composed of determined to need a forehead lift due to drooping upper eyelids (Experimental): The participant will visit the clinical trial institution at 4, 8, 12, and 16 weeks after the application visit (Visit 2, Baseline) of the medical device for clinical trials. They will participate in the efficacy evaluation of the clinical trial medical device for a total of 16 weeks.
  Interventions: Device: LinearZ

INTERVENTIONS:
Device: LinearZ — High Intensity Focues Ultrasound

SUMMARY:
Prospective, single center, single arm, open label study to evaluate the efficacy and safety of treatment with LinearFirm(ULTRAcel Q+) in temporary eyebrow lifting

DETAILED DESCRIPTION:
The goal of this open label study is to evaluate the efficacy and safety of treatment with HIFU system (LinearFirm(ULTRAcel Q+)) in temporary eyebrow lifting.

The target number of subjects for this clinical trial is set to 30 in a single group, without considering the statistical significance of hypothesis testing and dropout rate. Considering a dropout rate of 20%, the plan is to recruit a total of 38 subjects.

1. Evaluation of the effacacy is includes: Evaluation of eyebrow lifting photos by an independent evaluator, Patient Satisfaction (PS)
2. Evaluation of the safety is includes: Adverse events, vital signs, physical examination, and Visual Analogue Scale (VAS) after the application of medical devices for clinical trials

ELIGIBILITY:
Inclusion Criteria:

* 19 years old or older
* Voluntarily agreed to the clinical trial
* Who is need to eyebrow lifing

Exclusion Criteria:

* A history of cosmetic treatment (laser, light therapy, surgery, etc..) within the last 6 months
* A history of filler treatment (Collagen, AMA, etc...) within the last 6 months
* A history of Botulinum toxin injection within the last 6 months
* A history of treatment such as radiation therapy or chemotherapy, or history of malignat tumor
* A history of infections dermatitis, rash and shingles casued by thermal energy stimulation
* A history of treament with isotretinoin, retinoid preparations, or steroid preparations within the last 4 weeks
* Pregnancy
* Thos who participated in other clinical trials that affect the efficacy and safety evaluation of this clinical trial within 30 days of the screening date

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
The avegrage change in AEH (Average Eyebrow Height) and MEH(Maximum Eyebrow Height) compared to the Baseline | Base line and 4, 8, 12, 16weeks
  - Evaluation of the efficacy
  : Average change in AEH (Average Eyebrow Height) and MEH (Maximum Eyebrow Height) from the baseline, after the application of a medical device for clinical trials, as evaluated by an independent evaluator's eyebrow lifting photo evaluation at 4 weeks, 8 weeks, 12 weeks, and 16 weeks.
  This result will be displayed as a percentage.
The evaluation of the GLS (Glabellar Line Scale) compared to the Baseline | Base line and 4, 8, 12, 16weeks
  - Evaluation of the Exploratory
  1. The proportion of participants who showed an improvement of 2 points or more in the Glabellar Line Scale (GLS) evaluation of the most frowning state at 4 weeks, 8 weeks, 12 weeks, and 16 weeks after the application of a medical device for clinical trials, compared to the baseline.
  2. The proportion of participants who showed an improvement of 1 points or more in the Glabellar Line Scale (GLS) evaluation of the most frowning state at 4 weeks, 8 weeks, 12 weeks, and 16 weeks after the application of a medical device for clinical trials, compared to the baseline.
The evaluation of the TEAE (Treatment Emergent Adverse Event) and serious AE/ADE | after 16weeks
  1. The frequency and percentage of Treatment-Emergent Adverse Events (TEAE), Adverse Device Effects (ADE), and Serious Adverse Events/Adverse Device Effects (Serious AE/ADE) that occurred after the application of the medical device for clinical trials are presented.
  2. The frequency and percentage (%) of Treatment-Emergent Adverse Events (TEAE), Adverse Device Effects (ADE), and Serious Adverse Events/Adverse Device Effects (Serious AE/ADE) that occurred after the application of the medical device for clinical trials are presented.

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Sun, Study Director — Jeisys Medical Inc
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No